CLINICAL TRIAL: NCT06374914
Title: Sequential Intravesical Gemcitabine and Docetaxel for Rescue Therapy in BCG Unresponsive Non-muscle Invasive Bladder Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Muhammed Selcuk Ozer, Doctor, Dokuz Eylul University
Other Study IDs: TUO-UR-23-05
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer; BCG; Gemcitabine; Docetaxel; Intravesical Instillation
Keywords: bladder cancer; BCG; Intravesical Instillation; Gemcitabine; Docetaxel
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with BCG unresponsiveness and receiving intravesical gemcitabine doxetaxel
  Interventions: Drug: Intravesical Solution
- Patients with BCG unresponsiveness and radical cystectomy performed

INTERVENTIONS:
Drug: Intravesical Solution — Alkalinization of urine 1 day before the procedure Emptying the bladder with a catheter before the procedure mixing 1000 mg gemcitabine in 50 ml saline 90 minutes after administration 37.5 mg docetaxel mixed 120 minutes after administration in 50 ml saline maintanence if there is a 6 week induction response
  Other Names: Intravesical gemcitabin and docetaxel
  Groups: Patients with BCG unresponsiveness and receiving intravesical gemcitabine doxetaxel

SUMMARY:
Studies in the literature are limited both throughout Turkey and in general. For this reason, as a result of the study that we will create, it will provide us with information for bladder protective treatments in patients who do not respond to BCG therapy in bladder cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- BCG refractory/relapsed/unresponsive or intolerant Who do not want or are not suitable for radical cystectomy

Exclusion Criteria:

- BCG naive A history of multiple cancers Having a radical cystectomy plan

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a multi-center study within the scope of the Turkish Urooncology Association
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-09 (Estimated); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 5 years
  the recurrence rate after intravesical chemotherapy will be calculated
Progression rate | 5 years
  the progression rate after intravesical chemotherapy will be calculated
Adverse effects of intravesical chemotherapy | 5 years
  the patients' data will be retrospectively analyzed to investigate the side effects of intravesical chemotherapy
Intravesical chemotherapy versus radical cystectomy | 5 years
  the long-term cancer specific survival, overal survival, recurrence free survival of patients with similar pathological characteristics and who underwent radical cystectomy and patients who were given intravesical chemotherapy will be compared

SECONDARY OUTCOMES:
treatment change | 5 years
  patient transitions from intravesical chemotherapy to other treatment options will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Faculty of Medicine Department of Urology, Izmir, Other (Non U.s.), Turkey (Türkiye)